CLINICAL TRIAL: NCT06626347
Title: Application of the Telemedicine for Reach, Education, Access, and Treatment Delivery Model to Engage Emerging Adults in Diabetes Self-Management Education and Support
Brief Title: Telemedicine for Reach, Education, Access, and Treatment for Diabetes Self-Management Education and Support
Acronym: TREAT-ED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ingrid Libman, Associate Professor of Pediatrics and Epidemiology, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY24070160; R34DK136020 (NIH)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Type 1 Diabetes; Emerging Adults; Telemedicine; Health Care Delivery; Diabetes Self-Management Education and Support; Visit Attendance
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TREAT-ED (Experimental): * Emerging adult patients with type 1 diabetes assigned to groups of eight participants on average.
  * Four diabetes self-management education and support group sessions delivered virtually each session lasting 30-45 minutes.
  * Group sessions scheduled at intervals decided up on by participants.
  Interventions: Other: TREAT-ED Virtual Group Diabetes Self-Management Education and Support

INTERVENTIONS:
Other: TREAT-ED Virtual Group Diabetes Self-Management Education and Support — TREAT-ED is an innovative group telehealth delivery model designed to engage emerging adults in DSMES services. TREAT-ED sessions are facilitated by a Diabetes Care and Education Specialist and include content centered around the ADCES7 Self-Care Behaviors and applied learning strategies, e.g., case scenarios integrating glucose monitoring, and group discussions to drive knowledge transfer and skill development for diabetes self-care behaviors within the context of issues that are salient to the target population.

SUMMARY:
Emerging adults with type 1 diabetes are a vulnerable population. While diabetes self-management and education is known to offer opportunities to develop self-management skills required to achieve and maintain short- and long-term diabetes outcomes, emerging adults are reported to have poor clinic attendance and in turn low participation in diabetes self-management education and support services. This pilot study aims to test a novel approach to diabetes self-management education and support that incorporates technological and applied learning-driven methods delivered through group telemedicine visits to improve emerging adults engagement in diabetes self-management education and support with the ultimate goal of improving diabetes outcomes.

DETAILED DESCRIPTION:
Diabetes self-management education and support is considered a cornerstone of care and essential in helping people navigate self-management decisions and activities. Despite evidence that diabetes self-management education and support is a critical component of diabetes care, participation remains low. Emerging adulthood has been described as the distinct period between 18 and 25 years when adolescents work to achieve autonomy and explore life possibilities in moving toward adulthood. Suboptimal self-management has been identified as a major problem in emerging adults with type 1 diabetes, a particularly vulnerable group with an increased risk for poor diabetes-related outcomes. In its current form diabetes self-management education and support has been cited for not meeting the needs of emerging adults, when emerging adults have expressed interest in diabetes self-management education and support delivered with peer-supported, technological and applied learning-driven methods. To address these challenges, we are applying information gained from the literature and key stakeholder groups to our established Telemedicine for Reach, Education, Access and Treatment (TREAT) delivery model with a specific focus on diabetes self-management education and support. TREAT-ED (for self-management EDucation) will be designed to specifically engage emerging adults by integrating diabetes self-management education and support objectives to support informed decision making, self-care, and preparation for transfer to adult care, to improve outcomes. Diabetes care and education specialists will lead TREAT-ED with a cohort of emerging adults and will 1) help to organize and facilitate group sessions delivered through telehealth and 2) use continuous blood glucose monitoring reports as personalized examples to drive established diabetes self-management education and support content. With user-centered design techniques we developed and built and will now evaluate implementation determinants and test the TREAT-ED model. Feasibility assessment of the impact of the model on emerging adult patient participation in diabetes self-management education and support along with clinical, psychosocial and behavioral outcomes will be examined. We hypothesize that models that rely on current day strategies to engage emerging adults at high risk for diabetes-related problems with effective self-management skills will improve diabetes self-management education and support engagement and outcomes. If proven to be effective, this model is one that could be adapted for emerging adults who have transferred to adult diabetes care and other patient populations throughout the United States.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes (ICD10 E10.xx, O24.0x)
* 18 to 26 years of age at time of study enrollment
* Able to communicate via videoconferencing platform
* Intending to maintain status as a patient at participating clinical sites throughout the study duration
* Able to provide informed consent

Exclusion Criteria:

* Do not have a diagnosis of type 1 diabetes (ICD10 E10.xx, O24.0x)
* Less than 18 or older than 26 years old at time of enrollment
* Do not intend to maintain their care at participating clinical sites throughout the duration of the study
* Are unable to communicate via telemedicine
* Has other concerns that may interfere significantly with their ability to participate in the intervention (ongoing health issues, personal events, etc.)

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of diabetes self-management education and support sessions attended | From baseline to 6 months
  Possible range is 0 to 4 sessions.

SECONDARY OUTCOMES:
Change from baseline in empowerment at 6 months | Baseline vs. 6 months
  Empowerment will be assessed with the 8-item Diabetes Empowerment Scale-Short Form. Individual items are scored from 1 to 5; total scores are the average of all individual items. Higher scores indicate a greater sense of empowerment.
Change from baseline in readiness for transition at 6 months | Baseline vs. 6 months
  Transition readiness and self-management skill level will be assessed with the Transition Readiness Assessment Questionnaire. Individual items are scored from 1 to 5; total scores are the average of all individual items. The higher the score, the greater the readiness for transition to adult care.
Change from baseline in self-efficacy at 6 months | Baseline vs. 6 months
  Self-efficacy will be assessed using the 10-item Self-Efficacy for Diabetes Self-Management scale. Individuals items are scored from 1 to 10; total scores are the average of all individual items. Higher scores indicate greater self-efficacy.
Change from baseline in diabetes distress at 6 months | Baseline vs. 6 months
  Diabetes distress will be assessed with the Type 1 Diabetes Distress Assessment System: CORE SCALE. The CORE SCALE includes 8 items. Individual items are scored from 1 to 5; total scores are the average of all individual items. The higher the score, the greater the level of distress.
Change in percentage of patients with glycemic control from baseline to 6 months. | Baseline vs. 6 months
  Glycemic control defined as clinically measured hemoglobin A1c value of 7% or less. Values will be identified through medical record review.
Percentage of time in target glycemic range (70-180 mg/dL) | From baseline to 6 months
  Time in target glycemic range (70-180 mg/dL) is evaluated in 14 day periods using data recorded on continuous glucose monitoring systems and documented in the electronic health record system. This data will only be available for participants who use a continuous glucose monitor and provide data for documentation.
Number of acute care visits | From baseline to 6 months
  Number of emergency room visits and hospital admissions related to type 1 diabetes; documented in the medical record system.
Number of diabetes clinic visits attended | From baseline to 6 months
  Diabetes clinic visits with an endocrinologist are recommended to occur every three months or more frequently as needed at the participating institution and are documented in the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Libman, MD, PhD, Principal Investigator — University of Pittsburgh; Linda Siminerio, RN, PhD, CDCES, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD that underlies results reported in publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available after publication of primary results; available indefinitely.
Access Criteria: Investigators whose proposed research has received IRB approval will be able to access de-identified IPD that underlies published results, study protocol, SAP, and ICF.

DOCUMENTS (1):
  • Informed Consent Form (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT06626347/ICF_000.pdf